CLINICAL TRIAL: NCT06823271
Title: Haemodynamics and Ventricular Arrhythmias During Moderate-intensity Endurance and Resistance Exercise in Patients With Arrhythmogenic Cardiomyopathy, a Pilot Study
Brief Title: Haemodynamics and Ventricular Arrhythmias During Exercise in Patients With Arrhythmogenic Cardiomyopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-563-S-NP
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: In this interventional study patients will be separated into 2 groups with 10 patients per group Group 1: Patients with an implantable cardioverter-defibrillator Group 2: Patients without an implantable cardioverter-defibrillator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 with implantable cardioverter-defibrillator (Other): Patients with diagnosed definitive or borderline arrhythmogenic cardiomyopathy and implantable cardioverter-defibrillator will be included.
  Interventions: Other: Resting and exercise right heart catheterization; Other: Right ventricular mapping
- Group 2 without implantable cardioverter-defibrillator (Other): Patients with diagnosed definitive or borderline arrhythmogenic cardiomyopathy without implantable cardioverter-defibrillator will be included.
  Interventions: Other: Resting and exercise right heart catheterization; Other: Right ventricular mapping

INTERVENTIONS:
Other: Resting and exercise right heart catheterization — At rest and after different modes of exercise, exercise right heart catheterization will be performed.
Other: Right ventricular mapping — At the beginning and at the end of the exercise modes right ventricular mapping will be performed.

SUMMARY:
Patients with definitive and borderline arrhythmogenic cardiomyopathy (ACM) are usually recommended to refrain from high intensity exercise due to an increased risk of malignant arrhythmias. However, little is known about the effects of prolonged, low-to moderate endurance or resistance exercise on the burden of arrhythmias or central haemodynamics. This pilot interventional study assesses the impact of these modes of exercise on the electrophysiological substrate of the right ventricle (RV), measured by mapping of the RV, and central haemodynamics assessed by right heart catheterization. Patients older than 18 years of age with diagnosed borderline and definitive ACM are included with or without implantable cardioverter-defibrillator (ICD).

DETAILED DESCRIPTION:
This is a one-armed, monocentric, unblinded pilot interventional study. Upon fulfilment of the inclusion criteria (age >18 years of age, diagnosis of definitive or borderline ACM with or without implantable cardioverter defibrillator, ICD) and informed consent, patients will have two visits within one week.

The baseline exam (V1), consists of a clinical history, a questionnaire on the quality of life (Kansas City Cardiomyopathy Questionnaire, KCCQ), laboratory examination, echocardiography, 24h-Holter monitoring, and exertional cardiopulmonary exercise testing (CPET). Morphological (echocardiography) and functional (CPET) capacity of the participants will be assessed. With the aid of CPET, exercise intensity for continuous low to moderate-intensity endurance exercise during exercise right heart catheterization (exRHC) will be assessed (power at first ventilatory threshold). During V1 the one repetition maximum (1RPM) of isometric handgrip strength will be assessed as well as during dynamic flexion of the upper arm (biceps curl) with the contralateral arm of the planned venous puncture during the invasive testing.

Invasive Testing (V2): V2 will follow 48 hours after V1. Patients will first undergo supine resting right heart catheterization (RHC) followed by an electrophysiological study with mapping of the right ventricle (RV mapping) (condition 1, rest). Access for both procedures will be gained via the right internal jugular or brachial vein. After a 5-minute break isometric handgrip testing will assess haemodynamic changes (condition 2, isometric resistance test at 70% of the 1RPM for one minute). After another 5-minute break dynamic resistance testing will assess haemodynamic alterations (condition 3, dynamic resistance test, biceps curl at 70% of 1RPM for one minute with the contralateral arm of venous puncture). Following another 5-minute break, patients will perform supine bicycle exercise testing and haemodynamic measurements will be obtained at the end of 20 minutes of continuous, low to moderate-intensity endurance exercise (power at the first ventilatory threshold, condition 4, 20 minutes of moderate-intensity endurance test). Following haemodynamic testing, a prolonged low to moderate-intensity endurance exercise test will follow for another 20 minutes (power at the first ventilatory threshold), leading to a total time of 40 minutes, which is double the recommended duration from sports cardiology guidelines. Assessment of haemodynamics and RV mapping will be done at the end of this test (condition 5, 40-minutes low to moderate-intensity endurance test). In addition, cardiac biomarkers will be assessed before and after exercise.

Following invasive testing, patients without an ICD will receive an implantable loop recorder (ILR).

The aim of this interventional study is to assess changes of voltage maps during each of the exercise modes (20 minutes endurance test vs. 40 minutes endurance test vs. isometric handgrip vs. dynamic resistance exercise) as well as the change of pulmonary pressures. As patients with an ICD represent a high risk category, electrical and haemodynamic properties are compared between groups (ICD yes vs. no) in an exploratory approach. In this interventional study, which consists of assessments which are not part of routine medical care, the haemodynamic and electrophysiological effects of different exercise interventions (endurance and resistance tests) are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age
* Diagnosis of definitive or borderline arrhythmogenic cardiomyopathy (ACM) with or without implantable cardioverter defibrillator (ICD)

Exclusion Criteria:

* Age <18 years of age
* Manifest acute heart failure
* Intracardiac shunts
* Pre-existing precapillary pulmonary hypertension
* Clinical suspicion of new coronary artery disease or disease progression
* More than grade II valvular heart disease at resting echocardiography

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of the ratio of mean pulmonary artery pressure and cardiac output (mPAP/CO) between rest and the exercise tests in a patient | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Within each patient, the ratio of resting mean pulmonary artery pressure and cardiac output (mPAP/CO) will be compared to each exercise mode (isometric handgrip testing vs. dynamic resistance testing vs. 20minutes endurance exercise vs. 40 minutes endurance exercise) in a patient

SECONDARY OUTCOMES:
Difference of the pulmonary pulsatility index (PAPi) between rest and the exercise tests in a patient | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Within each patient, resting pulmonary pulsatility index (PAPi) will be compared to each exercise mode (isometric handgrip testing vs. dynamic resistance testing vs. 20minutes endurance exercise vs. 40 minutes endurance exercise) in a patient
Difference of the ratio of right atrial pressure to pulmonary artery wedge pressure (RA/PAWP) between rest and the exercise tests in a patient | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Within each patient, the ratio of resting right atrial pressure to pulmonary artery wedge pressure (RAP/PAWP) will be compared to each exercise mode (isometric handgrip testing vs. dynamic resistance testing vs. 20minutes endurance exercise vs. 40 minutes endurance exercise) in a patient
Difference of right ventricular power output reserve (RVPO reserve) between rest and exercise tests in a patient | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Right ventricular power output (RVPO) reserve (calculated as the difference between resting and exercise power output of the right ventricle (power output is calculated at rest and at the end of each condition as mean pulmonary artery pressure × cardiac output/451. Differences are compared within a patient between the exercise modes. Exercise modes are the following: Isometric handgrip testing vs. dynamic resistance testing vs. 20minutes endurance exercise vs. 40 minutes endurance exercise.
Change in voltage maps during resting and the different exercise modes per patient | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Voltage maps are compared in each patient between the resting measurement before exercise and after completion of all exercise modes (isometric handgrip testing, dynamic resistance testing, 20minutes endurance exercise, 40 minutes endurance exercise.)
Between group differences of the changes in the ratio of mean pulmonary artery pressure and cardiac output (mPAP/CO) between rest and the exercise tests | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Changes in the ratio of mean pulmonary artery pressure and cardiac output (mPAP/CO) between rest and the exercise modes will be compared between the two groups (patients with an implantable cardioverter defibrillator vs. those without). The exercise modes are the following: Isometric handgrip testing, dynamic resistance testing, 20minutes endurance exercise, 40 minutes endurance exercise.
Between group differences of the changes in voltage maps of the right ventricle between rest and the exercise tests. | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Changes in the voltage maps of the right ventricle (rest compared to the exercise modes) will be compared between the two groups (patients with an implantable cardioverter defibrillator vs. those without). The exercise modes are the following: Isometric handgrip testing, dynamic resistance testing, 20minutes endurance exercise, 40 minutes endurance exercise.
Between group difference of cardiac biomarkers etween rest and the exercise tests. | Through study completion, 48 hours after cardiopulmonary exercise testing (Visit 1)
  Changes in the cardiac biomarkers troponin I and N-terminal pro-B-type natriuretic peptide (rest compared to the exercise modes) will be compared between the two groups (patients with an implantable cardioverter defibrillator vs. those without). The exercise modes are the following: Isometric handgrip testing, dynamic resistance testing, 20minutes endurance exercise, 40 minutes endurance exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Wernhart, MD, Principal Investigator — Technical University Munich
Locations (1):
- Technische Universität München, München, Germany

IPD SHARING:
Plan to Share IPD: No
Individual data will only be shared anonymously on reasonable request to the principal investigator.

REFERENCES:
- [Result] Wernhart S, Goertz A, Hedderich J, Papathanasiou M, Hoffmann J, Rassaf T, Luedike P. Diastolic exercise stress testing in heart failure with preserved ejection fraction: The DEST-HF study. Eur J Heart Fail. 2023 Oct;25(10):1768-1780. doi: 10.1002/ejhf.2995. Epub 2023 Aug 24. PMID 37565370
- [Result] Gasperetti A, Rossi VA, Chiodini A, Casella M, Costa S, Akdis D, Buchel R, Deliniere A, Pruvot E, Gruner C, Carbucicchio C, Manka R, Dello Russo A, Tondo C, Brunckhorst C, Tanner F, Duru F, Saguner AM. Differentiating hereditary arrhythmogenic right ventricular cardiomyopathy from cardiac sarcoidosis fulfilling 2010 ARVC Task Force Criteria. Heart Rhythm. 2021 Feb;18(2):231-238. doi: 10.1016/j.hrthm.2020.09.015. Epub 2020 Sep 22. PMID 32976989
- [Result] Sawant AC, Te Riele AS, Tichnell C, Murray B, Bhonsale A, Tandri H, Judge DP, Calkins H, James CA. Safety of American Heart Association-recommended minimum exercise for desmosomal mutation carriers. Heart Rhythm. 2016 Jan;13(1):199-207. doi: 10.1016/j.hrthm.2015.08.035. Epub 2015 Aug 29. PMID 26321091
- [Result] Marcus FI, McKenna WJ, Sherrill D, Basso C, Bauce B, Bluemke DA, Calkins H, Corrado D, Cox MG, Daubert JP, Fontaine G, Gear K, Hauer R, Nava A, Picard MH, Protonotarios N, Saffitz JE, Sanborn DM, Steinberg JS, Tandri H, Thiene G, Towbin JA, Tsatsopoulou A, Wichter T, Zareba W. Diagnosis of arrhythmogenic right ventricular cardiomyopathy/dysplasia: proposed modification of the Task Force Criteria. Eur Heart J. 2010 Apr;31(7):806-14. doi: 10.1093/eurheartj/ehq025. Epub 2010 Feb 19. PMID 20172912
- [Result] Corrado D, Anastasakis A, Basso C, Bauce B, Blomstrom-Lundqvist C, Bucciarelli-Ducci C, Cipriani A, De Asmundis C, Gandjbakhch E, Jimenez-Jaimez J, Kharlap M, McKenna WJ, Monserrat L, Moon J, Pantazis A, Pelliccia A, Perazzolo Marra M, Pillichou K, Schulz-Menger J, Jurcut R, Seferovic P, Sharma S, Tfelt-Hansen J, Thiene G, Wichter T, Wilde A, Zorzi A. Proposed diagnostic criteria for arrhythmogenic cardiomyopathy: European Task Force consensus report. Int J Cardiol. 2024 Jan 15;395:131447. doi: 10.1016/j.ijcard.2023.131447. Epub 2023 Oct 14. PMID 37844667
- [Result] Cadrin-Tourigny J, Bosman LP, James CA. Sudden cardiac death risk prediction in arrhythmogenic right ventricular cardiomyopathy: a practical approach to navigating the challenges of prediction models. Eur Heart J. 2022 Dec 14;43(47):4961-4962. doi: 10.1093/eurheartj/ehac562. No abstract available. PMID 36263795
- [Result] Corrado D, Wichter T, Link MS, Hauer R, Marchlinski F, Anastasakis A, Bauce B, Basso C, Brunckhorst C, Tsatsopoulou A, Tandri H, Paul M, Schmied C, Pelliccia A, Duru F, Protonotarios N, Estes NA 3rd, McKenna WJ, Thiene G, Marcus FI, Calkins H. Treatment of arrhythmogenic right ventricular cardiomyopathy/dysplasia: an international task force consensus statement. Eur Heart J. 2015 Dec 7;36(46):3227-37. doi: 10.1093/eurheartj/ehv162. Epub 2015 Jul 27. No abstract available. PMID 26216920
- [Result] Saberniak J, Hasselberg NE, Borgquist R, Platonov PG, Sarvari SI, Smith HJ, Ribe M, Holst AG, Edvardsen T, Haugaa KH. Vigorous physical activity impairs myocardial function in patients with arrhythmogenic right ventricular cardiomyopathy and in mutation positive family members. Eur J Heart Fail. 2014 Dec;16(12):1337-44. doi: 10.1002/ejhf.181. Epub 2014 Oct 16. PMID 25319773